CLINICAL TRIAL: NCT03920982
Title: Determination of the Prognostic Value Serum Concentration of Indoxyl Sulfate During Acute Kidney Injury in Septic Shock Patients: TOX-AKI Study
Brief Title: Prognostic Value Serum Concentration of Indoxyl Sulfate During Acute Kidney Injury in Septic Shock Patients.
Acronym: TOX-AKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2018_843_0050
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Acute Kidney Injury; Septic Shock; Uremic; Toxemia; Mortality
Keywords: acute kidney injury; septic shock; uremic toxins; indoxyl sulfate; mortality
MeSH Terms: conditions — Acute Kidney Injury; Shock, Septic; Toxemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Determination of the blood concentration of indoxyl sulfate (IS) — IS concentration will be determined in blood of patients with septic shock and acute kidney injury. IS blood concentration will be done every day during 7 first days after patient will be admitted in intensive care unit. Relation between IS peak serum concentration and mortality at day 28 will be determined.

SUMMARY:
The development of acute kidney injury (AKI) during septic shock is frequent and is associated with a high mortality rate. The reason of this increased mortality despite the use of renal replacement therapy is still unknown. The deleterious effects of uremic toxins (solutes accumulating with the loss of kidney function) has risen for the last decade in chronic kidney disease patients. Among those solutes, indoxyl sulfate (IS) is associated with the development of cardiovascular complications and impairment of immune response. The role of uremic toxins and particularly IS in the prognostic of septic kidney injury is unknown. The investigators propose to analyze the relation between the serum concentration of IS and the mortality of patients hospitalized for a septic shock who developed an AKI.

DETAILED DESCRIPTION:
During chronic kidney disease the uremic toxins have been widely described as potential harmful solutes targeting the cardiovascular system, immunologic system, endothelium and bone metabolism. However, nothing is known about the potential accumulation and pejorative effects of those uremic toxins during AKI (Acute Kidney Injury). The objective of this study is to explore the role of the uremic toxins and specially IS (Indoxyl Sulfate) in the mortality of patients hospitalized for a septic shock and AKI. This study will also describe for the first time the kinetic of the blood concentration of different uremic toxins and their relation with the mortality and the kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years hospitalized in the medical intensive care unit in Amiens university hospital
* Presence of a septic shock (sepsis associated with a persistent hypotension after fluid resuscitation and requiring vasopressors to maintain MAP > 65 mmHg and/or serum lactate level > 2 mmol/ L).
* Evidence of AKI (KDIGO > or equal1) in the 72 hours following the admission in the ICU: diuresis < 0.5ml / kg / h for 6 to12 hours or > or equal 1.5 to1.9 fold increase or > 26.5 micromol / l in serum creatinine from baseline
* signed written informed consent form
* covered by national health insurance

Exclusion Criteria:

* known pre hospitalization (in the last 3 month preceding the hospitalization) advanced chronic kidney disease defined by an estimated glomerular filtration rate < 60 ml / min / 1.73m square
* Pregnancy
* Presence or strong clinical suspicion of renal obstruction
* Moribund patients (expected life < 48h)
* Cardio respiratory arrest
* Hemoglobin level below 10 g / dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Mortality rate | at day 28 after patient was admitted in intensive care unit
  Mortality of patients hospitalized for a septic shock who developed an acute kidney injury
Mortality rate | at day 90 after patient was admitted in intensive care unit
  Mortality of patients hospitalized for a septic shock who developed an acute kidney injury

SECONDARY OUTCOMES:
Blood concentration of indoxyl sulfate | at day 1 after patient was admitted in intensive care unit
  Blood concentration of indoxyl sulfate will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of indoxyl sulfate | at day 2 after patient was admitted in intensive care unit
  Blood concentration of indoxyl sulfate will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of indoxyl sulfate | at day 3 after patient was admitted in intensive care unit
  Blood concentration of indoxyl sulfate will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of indoxyl sulfate | at day 4 after patient was admitted in intensive care unit
  Blood concentration of indoxyl sulfate will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of indoxyl sulfate | at day 5 after patient was admitted in intensive care unit
  Blood concentration of indoxyl sulfate will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of indoxyl sulfate | at day 6 after patient was admitted in intensive care unit
  Blood concentration of indoxyl sulfate will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of indoxyl sulfate | at day 7 after patient was admitted in intensive care unit
  Blood concentration of indoxyl sulfate will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of para cresyl sulfate (PRS) | at day 1 after patient was admitted in intensive care unit
  Blood concentration of para cresyl sulfate (PRS) will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of para cresyl sulfate (PRS) | at day 2 after patient was admitted in intensive care unit
  Blood concentration of para cresyl sulfate (PRS) will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of para cresyl sulfate (PRS) | at day 3 after patient was admitted in intensive care unit
  Blood concentration of para cresyl sulfate (PRS) will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of para cresyl sulfate (PRS) | at day 4 after patient was admitted in intensive care unit
  Blood concentration of para cresyl sulfate (PRS) will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of para cresyl sulfate (PRS) | at day 5 after patient was admitted in intensive care unit
  Blood concentration of para cresyl sulfate (PRS) will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of para cresyl sulfate (PRS) | at day 6 after patient was admitted in intensive care unit
  Blood concentration of para cresyl sulfate (PRS) will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of para cresyl sulfate (PRS) | at day 7 after patient was admitted in intensive care unit
  Blood concentration of para cresyl sulfate (PRS) will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of FGF 23 (Fibroblast Growth Factor 23) | at day 1 after patient was admitted in intensive care unit
  Blood concentration of FGF 23 (Fibroblast Growth Factor 23) will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of FGF 23 (Fibroblast Growth Factor 23) | at day 2 after patient was admitted in intensive care unit
  Blood concentration of FGF 23 (Fibroblast Growth Factor 23) will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of FGF 23 (Fibroblast Growth Factor 23) | at day 3 after patient was admitted in intensive care unit
  Blood concentration of FGF 23 (Fibroblast Growth Factor 23) will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of FGF 23 (Fibroblast Growth Factor 23) | at day 4 after patient was admitted in intensive care unit
  Blood concentration of FGF 23 (Fibroblast Growth Factor 23) will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of FGF 23 (Fibroblast Growth Factor 23) | at day 5 after patient was admitted in intensive care unit
  Blood concentration of FGF 23 (Fibroblast Growth Factor 23) will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of FGF 23 (Fibroblast Growth Factor 23) | at day 6 after patient was admitted in intensive care unit
  Blood concentration of FGF 23 (Fibroblast Growth Factor 23) will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of FGF 23 (Fibroblast Growth Factor 23) | at day 7 after patient was admitted in intensive care unit
  Blood concentration of FGF 23 (Fibroblast Growth Factor 23) will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of Klotho | at day 1 after patient was admitted in intensive care unit
  Blood concentration of Klotho will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of Klotho | at day 2 after patient was admitted in intensive care unit
  Blood concentration of Klotho will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of Klotho | at day 3 after patient was admitted in intensive care unit
  Blood concentration of Klotho will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of Klotho | at day 4 after patient was admitted in intensive care unit
  Blood concentration of Klotho will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of Klotho | at day 5 after patient was admitted in intensive care unit
  Blood concentration of Klotho will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of Klotho | at day 6 after patient was admitted in intensive care unit
  Blood concentration of Klotho will be measured in patients hospitalized for a septic shock who developed an acute kidney injury
Blood concentration of Klotho | at day 7 after patient was admitted in intensive care unit
  Blood concentration of Klotho will be measured in patients hospitalized for a septic shock who developed an acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: michel slama, Pr, Principal Investigator — CHU Amiens; Clement Brautt, MD, Principal Investigator — CHU Amiens; Yoan Zerbib, MD, Principal Investigator — CHU Amiens; Youssef Bennis, Dr, Principal Investigator — CHU Amiens; Sandra Bodeau, Dr, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No